CLINICAL TRIAL: NCT04419636
Title: Interventional, Open-label, Position Emission Tomography (PET) Study Investigating MAGL Occupancy After Single and Multiple Oral Doses of Lu AG06466 in Healthy Male Subjects
Brief Title: Binding of Lu AG06466 in the Brain in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18454A
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Healthy
MeSH Terms: interventions — ABX-1431

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A Single doses (Experimental): Lu AG06466 in fast and fed state
  Interventions: Drug: Lu AG06466
- Part B Repeated doses (Experimental): Lu AG06466 after light meal
  Interventions: Drug: Lu AG06466

INTERVENTIONS:
Drug: Lu AG06466 — capsules, orally
  Other Names: ABX-1431

SUMMARY:
A study to learn how Lu AG06466 and one of its break down products binds in the brain after single and repeated dosing

DETAILED DESCRIPTION:
The study will be conducted in two Parts. Part A: cross over, fed/fasted determined by randomized sequence Part B: sequential group

PET scans will be used to quantify MAGL occupancy

ELIGIBILITY:
Inclusion Criteria:

* body weight ≥60 kg.
* body mass index ≥18.5 and ≤27 kg/m2.
* waist circumference ≤94 cm.
* The subject has a normal sMRI performed during the screening period.
* The subject is suitable for radial artery blood sampling and cannulation as demonstrated by the Allen test.
* Subject must be healthy as assessed using detailed medical history, laboratory tests, and physical examination.
* The subject must make use of contraception.

Exclusion Criteria:

* The subject is left handed.

Other in- and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Central monoacylglycerol lipase (MAGL) occupancy | From dosing to 8 hours post-dose

SECONDARY OUTCOMES:
C(PET) | From zero to Day 10
  Average plasma concentration for Lu AG06466 and Lu AG06988 during PET imaging
AUC (0-24) | From zero to 24 hours post-dose
  Area under the plasma concentration curve for Lu AG06466 and Lu AG06988 from zero to 24 hours
Cmax | From zero to 24 hours post-dose
  Maximum observed plasma concentration for Lu AG06466 and Lu AG06988

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- UZ Leuven campus Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided